CLINICAL TRIAL: NCT04401761
Title: Xarelto + Acetylsalicylic Acid: Treatment Patterns and Outcomes Across the Disease Continuum in Patients With CAD and/or PAD
Brief Title: A Study to Collect Data on the Treatment Pattern of Xarelto + Acetylsalicylic Acid in the Routine Clinical Practice in Patients Who Are Suffering From a Condition That Narrows the Blood Vessels Supplying the Heart and / or a Condition That Most Commonly Narrows the Blood Vessel in the Legs
Acronym: XATOC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21283
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Peripheral Artery Disease
Keywords: Thrombosis
MeSH Terms: conditions — Coronary Artery Disease; Peripheral Arterial Disease; Thrombosis | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAD/PAD-patients: Adult patients with coronary artery disease (CAD) or symptomatic peripheral artery disease (PAD) who are treated with a combination of rivaroxaban and acetylsalicylic acid.
  Interventions: Drug: Rivaroxaban (BAY59-7939, Xarelto); Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939, Xarelto) — 2.5 mg twice daily
  Other Names: Xarelto
Drug: Acetylsalicylic acid — 75 - 100 mg once daily at the discretion of the investigator
  Other Names: Aspirin

SUMMARY:
The study will focus on effectiveness and safety of rivaroxaban (Xarelto) when given together with acetylsalicylic acid (combination therapy) to patients suffering from coronary artery disease (a condition that affects the blood vessels supplying the heart) and / or peripheral artery disease (a condition that affects the blood vessels of the lower limbs) in the routine clinical practice. The study will help to collect data for prevention cardiovascular death, myocardial infarction (MI), stroke and major adverse limb events in adult patients. The study will focus on information on when and why physicians are starting to treat patients with combination therapy, treatment duration, reasons to discontinue treatment and previous therapies. The study will also investigate treatment outcomes for patients being treated with a combination therapy by their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patient (except Taiwan ≥ 20 years old).
* Diagnosis of CAD or symptomatic PAD.
* Treatment according to local marketing authorization, rivaroxaban 2.5 mg [BID] plus Acetylsalicylic acid (ASA) 75-100 mg [OD] started up to 4 weeks before or after the ICF is signed.
* Only in those countries with a marketing authorization of rivaroxaban in the Acute Coronary Syndrome (ACS) indication, patients already on rivaroxaban treatment for ACS for more than 4 weeks, who are subsequently fulfilling criteria for CAD, are also allowed to be enrolled.

Exclusion Criteria:

* Contra-indications according to the local marketing authorization.
* Patients who will be treated with chronic anticoagulation therapy other than rivaroxaban 2.5 mg given for CAD/PAD.
* Participation in an interventional trial.
* Enrolment in the XATOA study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: International population of adult CAD/PAD patients
Sampling Method: Non-Probability Sample
Enrollment: 3189 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Health status by questionnaire EQ-5D-5L | Up to 34 months
  Self-reported health-related quality of life is measured with EQ-5D at the initial visit and at each follow-up visit. Items are scored from 1 (no problems) to 5 (extreme problems) leading to a total score from 0 (worst imaginable health) to 100 (best imaginable health).
Descriptive analysis of clinical characteristics of CAD participants | At baseline
Descriptive analysis of clinical characteristics of PAD participants | At baseline
Descriptive analysis of prior antithrombotic treatment | At baseline
Descriptive analysis of concomitant antithrombotic treatment | Upto 34 months
Descriptive analysis of prior secondary prevention therapies | At baseline
Descriptive analysis of concomitant secondary prevention therapies | Up to 34 months
Reason to start rivaroxaban | At baseline
  Reasons include past ischemic events, co-morbidities and medical history.
Decision point to start rivaroxaban | At baseline
  Time point of start of medication in relation to disease progress and/ or occurrence of ischemic events
Reasons for discontinuation of rivaroxaban | Up to 34 months
Planned duration of treatment with rivaroxaban | At baseline
Actual duration of treatment with rivaroxaban | Up to 34 months
Planned duration of treatment with Acetylsalicylic acid (ASA) | At baseline
Actual duration of treatment with ASA | Up to 34 months

SECONDARY OUTCOMES:
Number of participants with major adverse cardiovascular events (MACE) | Up to 34 months
  Composite endpoint comprising of myocardial infarction, stroke, and cardiovascular death (and single components).
Number of participants with major adverse limb events (MALE) | Up to 34 months
  Major adverse limb events comprise acute limb ischemia and vascular amputation, and antithrombotic treatment [pattern] after MALE.
Number of participants with antithrombotic treatment after MALE | Up to 34 months
Number of participants with MACE or MALE | Up to 34 months
  Composite endpoint comprising myocardial infarction, ischemic stroke, cardiovascular death, acute limb ischemia, major amputation of vascular etiology.
Number of participants with thromboembolic events | Up to 34 months
  Thromboembolic events include e.g. systemic embolism and venous thromboembolism.
Number of participants with haemorrhagic events and complications | Up to 34 months
  The major bleeding complications will be collected according to the International Society on Thrombosis and Haemostasis (ISTH) criteria, modified ISTH criteria, and Thrombolysis in Myocardial Infarction (TIMI) criteria.
Number of deaths due to cardiovascular events | Up to 34 months
Number of deaths due to any cause | Up to 34 months
Number of participants with cardiac revascularization procedures | Up to 34 months
  Cardiac revascularization procedure includes Percutaneous Coronary Intervention (PCI), Coronary Artery Bypass Grafting (CABG)
Number of participants with peripheral revascularization procedures | Up to 34 months
Number of participants with lower limb revascularization procedures. | Up to 34 months
Number of participants with carotid revascularization procedures | Up to 34 months
Number of hospitalizations | Up to 34 months
  Number of hospitalizations due to stroke, cardiovascular reasons, MALE, or bleeding complications.
Duration of hospitalizations | Up to 34 months
  Hospitalizations due to stroke, cardiovascular reasons, MALE, or bleeding complications.
Total walking distance per individual for PAD participants | Up to 34 months
Pain free walking distance per individual for PAD participants | Up to 34 months
Patient-reported walking impairment by Walking Impairment Questionnaire (WIQ) for PAD participants | Up to 34 months
  The WIQ is a validated questionnaire that measures patient-reported walking limitations in distance, stair climbing and speed. Final score ranges from 0 (unable to walk) to 4 (no difficulty to walk).

CONTACTS AND LOCATIONS:
Locations (10):
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Colombia
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Slovenia
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.